CLINICAL TRIAL: NCT04459325
Title: A Prospective Open-label Study of the Tigerase® Efficacy and Safety as Part of Complex Therapy in Patients With COVID-19
Brief Title: Tigerase® Efficacy and Safety as Part of Complex Therapy in Patients With COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AO GENERIUM (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DRN-ALI-III; #216 eff date 27.05.2020 (Other: Ministry of Health of Russia)
Record Dates: First submitted 2020-07-03; First posted 2020-07-07 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-07

CONDITIONS: COVID-19; Coronavirus Disease 2019
Keywords: COVID-19; Coronavirus Infections; Coronaviridae Infections; Dornase alfa; Virus Diseases; Acute lung injury; Acute respiratory distress syndrome; Respiratory Insufficiency; Respiratory Tract Diseases
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Coronaviridae Infections; Virus Diseases; Acute Lung Injury; Respiratory Distress Syndrome; Respiratory Insufficiency; Respiratory Tract Diseases | interventions — dornase alfa; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study drug and best available care (Experimental): Best available care and Tigerase®/nebulised dornase alfa [2.5 mg BID] for 7 days
  Interventions: Biological: Tigerase® and best available care
- Control group (best available care) (Other): Patients will receive the usual care in accordance with good practice.
  Interventions: Other: Best available care

INTERVENTIONS:
Biological: Tigerase® and best available care — Nebulised dornase alfa [2.5 mg BID] for 7 days
  Other Names: Dornase Alfa Inhalation Solution and best available care
  Arms: Study drug and best available care
Other: Best available care — Patients will receive the usual care in accordance with good practice.
  Other Names: Standard of care
  Arms: Control group (best available care)

SUMMARY:
It is a multicenter, open-label, randomized, parallel-group study of the efficacy and safety of Tigerase® (GENERIUM JSC, Russia) with standard therapy versus standard therapy in patients with COVID-19.

DETAILED DESCRIPTION:
COVID-19 (Coronavirus disease-19) is an acute respiratory infectious disease caused by SARS-CoV-2 coronavirus. The spread of the disease quickly developed to the global pandemic in March-April 2020, and was characterized by acute respiratory distress syndrome (ARDS) in 10-15% of cases, which leads to a high frequency of hospitalization in the intensive care unit and high mortality. The search for effective treatment and reducing the severity of COVID-19 is a priority in the development of medical science.

One of the key processes of the innate immune system are neutrophil extracellular traps (NET), formed by neutrophils when they eject their DNA from the cytoplasm. NET is most often described as a mechanism for capturing bacteria in order to limit their spread. In addition, NET also plays a role in antiviral immunity. In particular, viral infections lung damage is at least partially due to NET.

This suggests that drug disruption of NET in COVID-19 is promising. DNase preparations, and in particular Tigerase®, are safe and effective for the treatment of cystic fibrosis and can serve as a NET destruction agent in patient with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent for participation in the study
2. Men and women aged ≥18 years
3. Laboratory-confirmed diagnosis of coronavirus infection caused by COVID19, moderate severity *

   *Criteria for moderate flow (just one point) Mandatory Criterion
   * Pneumonia Additional criteria (used to characterize the disease and are not required to determine the severity)
   * Fever above 38 ° C
   * respiratory rate more than 22 / min
   * Shortness of breath during physical exertion
   * SpO2 <95%
   * С-reactive protein (CRP) of serum more than 10 mg / l
4. Patients with pneumonia with a stable level of hemoglobin saturation by oxygen (> 93%) on oxygen support and / or receiving respiratory support of non-invasive mechanical ventilation

Exclusion Criteria:

1. Individual intolerance or hypersensitivity to the active or any of the excipients of the drug Tigerase®
2. The need for invasive mechanical ventilation at the time of inclusion of the patient
3. Patients severe condition (one of the following characteristics):

   * Respiratory distress syndrome with respiratory rate ≥30 per minute
   * Saturation of hemoglobin with oxygen ≤93% with oxygen support
4. Patient participate in any clinical trials and / or taking the experimental drug within 30 days before inclusion this trial
5. Severe competitive respiratory system diseases (bronchial asthma, chronic obstructive pulmonary disease - COPD, cystic fibrosis, interstitial lung disease)
6. Positive results of laboratory testing for HIV and hepatitis B and C
7. Life expectancy less than 12 months without COVID-19
8. Other diseases and conditions, significant laboratory or instrumental deviation, which, according to investigator opinion, may impact the results of the study, limit the patient's participation in the trial or create an unreasonable risk for the patient
9. Patient's unwillingness or disability to comply with the recommendations prescribed by protocol, as well as any concomitant medical or serious mental conditions that render the patient unsuitable for participation in the study, limit the legitimacy of obtaining informed consent or may affect the patient's ability to participate in the study (including disability to use a nebulizer)
10. Positive pregnancy test in women
11. The period of breastfeeding in women
12. Refusal of male patients and female patients with preserved reproductive function to use adequate methods of contraception throughout the study and for at least 30 days after the end of therapy with the studied drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with mechanical ventilation | Day 8
Category change on WHO Ordinal Scale for Clinical Improvement | Day 8

SECONDARY OUTCOMES:
The proportion of patients with mechanical ventilation | Day 28
Category change on WHO Ordinal Scale for Clinical Improvement | Day 28
Proportion of patients surviving 28 days after inclusion in the study | Day 28
Number of days of oxygen therapy during the treatment period | Day 8
Change in C-reactive protein level | Days 3, 5, 8
Change in oxygenation index | Days 3, 5, 8
  PaO2 / FiO2, FiO2 = fraction of oxygen in inhaled air,% PaO2 = partial pressure of oxygen in arterial blood, mm Hg
Change in SpO2/FiO2 index | Days 1, 2, 3, 4, 5, 6, 7, 8
  SpO2 / FiO2, FiO2 = fraction of oxygen in inhaled air,% SpO2 = hemoglobin oxygen saturation, %
Change in ferritin level | Days 3, 5, 8
Change in D-dimer level | Days 3, 5, 8
Change in neutrophil-leucocyte ratio | Days 3, 5, 8
Change in leucocyte-C-reactive protein ratio | Days 3, 5, 8
Change in the level of relative (%) number of lymphocytes of the general blood test | Days 3, 5, 8

CONTACTS AND LOCATIONS:
Overall Officials: Oksana A. Markova, MD, Study Chair — AO GENERIUM
Locations (6):
- Russia (6):
  - City Clinical Hospital #15, Moscow
  - I.M. Sechenov First Moscow State Medical University (Sechenov University), Moscow
  - City Clinical Hospital #51, Moscow
  - City Clinical Hospital #52, Moscow
  - N.V. Sklifosovsky Scientific Research Institute of First Aid, Moscow
  - Siberian State Medical University (SibMed), Moscow

IPD SHARING:
Plan to Share IPD: No